CLINICAL TRIAL: NCT06029764
Title: Extended One-level Interbody Fusion for Adjacent Vacuum Phenomenon in Lumbar Degenerative Disc Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuASD
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Adjacent Segment Degeneration

STUDY DESIGN:
Intervention Model Description: This study will use a simple randomization method to group patients who meet the inclusion criteria using a computer-generated randomization scheme.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The study will enroll patients with lumbar degeneration undergoing 1-2 level intervertebral fusion, and for patients with asymptomatic and non-instability intervertebral discs adjacent to the operative level with vacuum signs, extended one-level interbody fusion will be performed.
  Interventions: Procedure: extended one-level interbody fusion
- control group (No Intervention): The control group underwent intervertebral fusion only at the responsible segment.

INTERVENTIONS:
Procedure: extended one-level interbody fusion — For patients who have vacuum signs in the intervertebral disc adjacent to the surgical segment but are asymptomatic and not unstable, the intervertebral fusion surgery is extended to one segment and followed up immediately after surgery, 3 months, 6 months, and annually within 1 to 5 years. Take lumbar spine MR to determine the degree of degeneration progression of adjacent segments and whether revision surgery is needed. Take X-rays of the lumbar spine in frontal and lateral + flexion and extension positions, and CT-three-dimensional reconstruction to judge the bony fusion of the intervertebral fusion.
  Arms: experimental group

SUMMARY:
The main objective of this study was to validate the clinical effectiveness of interbody fusion with a one-segment extension for the treatment of adjacent segmental space discs in the surgical treatment of lumbar degeneration.

DETAILED DESCRIPTION:
The study will include patients with lumbar degeneration who underwent 1-2 segment interbody fusion, and for patients with vacuum signs but no symptoms and no instability of the discs in the adjacent segments of the operated segments, lumbar interbody fusion will be extended by one segment, and the patients will be followed up annually in the immediate postoperative period, in March, June, and in the period of 1-5 years, and lumbar MR will be taken at the time of follow-up to determine the degree of progression of the degeneration in the neighboring segments, and whether or not revision surgery is needed. The lumbar spine was photographed in the frontal and lateral + anterior flexion and posterior extension X-rays and CT-3D reconstruction to determine the bony fusion of the interbody fusion. In addition, the lumbar spine ODI score was applied for evaluation at the follow-up visit, and the total lumbar spine-related expenses of the patients up to the follow-up visit were recorded.

ELIGIBILITY:
Inclusion Criteria:

* The age was between 18-60 years old; patients with lumbar degeneration required 1-2 segment interbody fusion, and there were vacuum signs but no symptoms and no instability of the discs in the adjacent segments (power position slip ≤3mm and segmental angle change ≤10°); they agreed with the surgical plan and were willing to undergo long-term clinical follow-up, and signed an informed consent form.

Exclusion Criteria:

* Drug or alcohol abusers; those with abnormal liver or kidney function unsuitable for surgery; those with cardiac insufficiency unsuitable for surgery; those with severe metabolic and endocrine diseases unsuitable for surgery; those with severe lung disorders such as asthma and abnormal lung function unsuitable for surgery; pregnant and breastfeeding women as well as those who are planning to become pregnant in the near future; those who have participated in other clinical trials within 3 months; and those who are not suitable for participation in the experiment in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Surgical revision rate | Postoperative month 3 (±15 days), month 6 (±15 days), yearly for 5 years (±30 days)
  MR of the lumbar spine was taken at follow-up to determine the degree of progression of degeneration in the neighboring segments and the need for revision surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fengzeng Jian, MD,PhD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kanna RM, Hajare S, Thippeswamy PB, Shetty AP, Rajasekaran S. Advanced disc degeneration, bi-planar instability and pathways of peri-discal gas suffusion contribute to pathogenesis of intradiscal vacuum phenomenon. Eur Spine J. 2022 Mar;31(3):755-763. doi: 10.1007/s00586-022-07122-0. Epub 2022 Jan 28. PMID 35089418
- [Result] Wang T, Ding W. Risk factors for adjacent segment degeneration after posterior lumbar fusion surgery in treatment for degenerative lumbar disorders: a meta-analysis. J Orthop Surg Res. 2020 Dec 3;15(1):582. doi: 10.1186/s13018-020-02032-7. PMID 33272288
- [Result] Ghiselli G, Wang JC, Bhatia NN, Hsu WK, Dawson EG. Adjacent segment degeneration in the lumbar spine. J Bone Joint Surg Am. 2004 Jul;86(7):1497-503. doi: 10.2106/00004623-200407000-00020. PMID 15252099